CLINICAL TRIAL: NCT06390904
Title: Gonadotropin-releasing Hormone Agonist (GnRHa) Plus Letrozole in Obese Progestin-insensitive Endometrial Atypical Hyperplasia Patients With Conservative Treatment
Brief Title: GnRHa + Letrozole in Obese Progestin-insensitive Endometrial Atypical Hyperplasia Patients
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Xiaojun Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaojun Chen, Professor, Fudan University
Organization: Fudan University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 53211030-3
Record Dates: First submitted 2024-04-22; First posted 2024-04-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Atypical Endometrial Hyperplasia; Progesterone Resistance; Obesity
MeSH Terms: conditions — Endometrial Hyperplasia; Progesterone Resistance; Obesity | interventions — LHRH, Ac-Nal(1)-Cpa(2)-Trp(3)-Arg(6)-Ala(10)-; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Obese EAH group (Experimental): This group including 29 EAH cases. Interventional Study Model was Simon two-stage optimal design. Eleven patients were needed for the first stage, and if eight or more patients achieved CR at 28 weeks, the trial can enter into the second stage.
  Then every 12 to 16 weeks, an hysteroscope will be used to evaluate the endometrial condition, and the pathological findings will be recorded.
  Interventions: Drug: GnRH antagonist; Drug: Letrozole 2.5mg

INTERVENTIONS:
Drug: GnRH antagonist — Gonadotropin-releasing hormone analogue, intramuscular injection of 3.75mg will be given every 4 weeks, and the maximum treatment courses will be 6. If the patient get CR within 6 courses, another 2 courses will be used as consolidation therapy.
Drug: Letrozole 2.5mg — 2.5mg po qd.

SUMMARY:
To investigate the efficacy of Gonadotropin-releasing Hormone Agonist (GnRHa) plus letrozole in obese progestin-insensitive atypical endometrial hyperplasia (EAH) patients.

DETAILED DESCRIPTION:
There were more and more women with early endometrioid endometrial cancer (EEC) and atypical endometrial hyperplasia (EAH) who want to preserve fertility.

Approximately 70% to 80% of females who meet the criteria for conservation treatment are able to achieve complete response (CR) after progestin therapy, with a median time of 6-7 months, but about 20% to 30% of patients get no response or need to take longer time to achieve remission (over one year). With long duration of treatment, there will be more side effects such as weight gain, impaired liver function, endometrial injury, ovarian reserve inhibition etc. which will decrease the efficacy of conservative treatment. Previous researches had shown that Gonadotropin-releasing Hormone Agonist (GnRHa) plus letrozole could be a better second-line treatment for obese progestin-insensitive patients. Till now, no similar studies were found, so the investigators design this study to explore the efficacy of GnRHa plus letrozole in obese progestin-insensitive EAH patients to provide new evidences for improving conservative treatment efficacy. The investigators defined obese patients as these with BMI ≥ 30kg/m^2.

This will be a single-centred prospective pilot study. Patients diagnosed as obese progestin-insensitive EAH by dilatation and curettage (D&C) or hysteroscopy will be enrolled. The primary endpoint is cumulative CR rate at 28 weeks of treatment. The secondary endpoints include adverse events, duration of complete response, recurrent rate, pregnancy rate and quality of life of patients.

ELIGIBILITY:
Inclusion Criteria:

* Have a confirmed initial pathological diagnosis based upon hysteroscopy: histologically prove EAH
* BMI≥30kg/m2
* Using progestin, any of the following therapy, as first-line treatment:

  1. Megestrol acetate ≥ 160 mg qd using, combined with Levonorgestrel Lntrauterine System (LNG-IUS) inserted or not
  2. Medroxyprogesterone acetate ≥ 250 mg qd using, combined with LNG-IUS inserted or not
  3. LNG-IUS inserted
* Progestin-insensitive:

  1. remained with stable disease after 7 months of progestin use
  2. did not achieve CR after 10 months of progestin use
* Have a desire for remaining reproductive function or uterus
* Good compliance with adjunctive treatment and follow-up

Exclusion Criteria:

* Combined with severe medical disease or severely impaired liver and kidney function
* Pathologically confirmed as endometrial cancer with suspicious myometrial invasion or extrauterine metastasis
* Patients with other types of endometrial cancer or other malignant tumors of the reproductive system
* Patients with breast cancer or other hormone- dependent tumors or diseases that cannot be used with GnRHa or Letrozole
* Strong request for uterine removal or other conservative treatment
* Known or suspected pregnancy
* Acute severe disease such as stroke or heart infarction or a history of thrombosis disease
* Smoker(>15 cigarettes a day)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Estimated)
Dates: Start 2022-07-13 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) rate within 28 weeks of treatment | Up to 28 weeks
  The cumulative 28-week CR rate will be calculated. Patients will be evaluated with an hysteroscopy every 12 to 16 weeks. The response to progestin treatment was assessed histologically using specimens obtained during each hysteroscopic evaluation. CR was defined as the absence of hyperplasia or carcinoma.

SECONDARY OUTCOMES:
Adverse events | During the treatment period, an average of 28 weeks
  Adverse effects were recorded during the entire treatment period, including weight gain, thrombosis, lactic acidosis, abnormal liver and renal function, and other toxicities or complaints.
Time to achieve CR | During the treatment period, an average of 28 weeks
  The median CR time will be calculated.
Relapse rate | Average of 2 years after the completion of the treatment
  Relapse will be defined as endometrial hyperplasia or endometrial cancer recurred after patients achieve CR.
Rate of fertility outcomes | Average of 2 years after the completion of the treatment
  Among patients prepared to get pregnant, fertility outcomes will be recorded.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tenth People's Hospital of Tongji University, Shanghai, Shanghai Municipality
  - Obstetrics and Gynecology Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhou S, Xu Z, Yang B, Guan J, Shan W, Shi Y, Chen X. Characteristics of progestin-insensitive early stage endometrial cancer and atypical hyperplasia patients receiving second-line fertility-sparing treatment. J Gynecol Oncol. 2021 Jul;32(4):e57. doi: 10.3802/jgo.2021.32.e57. PMID 34085795